CLINICAL TRIAL: NCT04482764
Title: The Effectiveness of Valproic Acid in Treating Frequent Cyanotic Breath Holding Spells
Brief Title: Valproic Acid in Treating Cyanotic Breath Holding Spells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherifa Ahmed Hamed, Professor of Neurology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-VPA-SH-2017
Record Dates: First submitted 2017-10-03; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Breathhold
Keywords: Breath holding spells; cyanosis; valproic acid
MeSH Terms: conditions — Cyanosis | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cyanotic breath holding spells (Other): drug, valproic acid: 5mg/kg/d for 6 months
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — Treatment of children with frequent cyanotic breath holding spells (at least 4 spells per week) with 5 mg/kg/day for 6 months.
  Other Names: sodium valproate

SUMMARY:
Breath holding spells (BHS) are common non-epileptic paroxysmal behavioral involuntary episodes occurring in up to 5.9% of healthy children. The attacks occur in early childhood (0.5-3 years) but are self-limited by school age (4-5 years old) (90%). Classically, BHS were classified as cyanotic (blue), pallid (pale) and mixed based on the color change of the child during the spell. In general, cyanotic spells have been classically described in a toddler with excessive temper tantrums [stubborn, easily frustration or annoyed. The mechanisms of BHS are controversial. The most suggested cause of BHS is instability of the autonomic nervous system, inhibition of respiratory effort and cyanosis in cyanotic BHS and bradycardia or a brief asystole and cerebral hypoperfusion in pallid BHS. Iron deficiency anemia (IDA) has been widely regarded as a risk factor for BHS in nearly 50% of children due to reduced brain oxygenation [4]. It is generally agreed that the long-term prognosis is considered good [1]. There is no definite therapy for BHS. In children with low frequency spells, parental reassurance are just enough; however, high frequency spells may result in anxiety to the parents or fear from sudden death of the child or development of mental subnormality. Treatment of iron has been reported to result in reduction of the frequency of spells or its stoppage. Some reported improvement of BHS with piracetam [a nootropic drug known to increase brain oxygenation]. We did not find systematized published reports evaluating the effectiveness of antiepileptic drugs (AEDs) in reduction of spells frequency of cyanotic BHS or their stoppage.

ELIGIBILITY:
Inclusion criteria :

1. Children with high frequency spells (≥ 4/week) of CBHS.
2. Children with parents who were wishing to provide treatment to their children.
3. Failure of alternatives modalities of treatment (e.g. iron supplements, piracetam, non-specific vitamins, etc) (tried for ≥ 3 months) to reduce the frequency of spells or stop them.
4. Follow-up for 6 months after starting treatment with valproic acid.

Exclusion criteria:

1. Primary neurologic disease, history of epilepsy or febrile convulsions, abnormal neurological examination and abnormal EEG.
2. Primary cardiac disease or presence of long QT syndrome in the ECG.
3. Presence of a hematologic (other than IDA) or other medical disease, electrolyte disturbance, hypoglycemia, hypocalcemia, impaired kidney or liver function tests.
4. Those with a doubtful diagnosis.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
frequency of spells after starting treatment with valproic acid | 6 months
  The parents or legal guardians are the sources of information about the frequency of spells.

CONTACTS AND LOCATIONS:
Overall Officials: Sherifa A Hamed, M.D., Principal Investigator — Assiut University, Faculty of Medicine
Locations (1):
- Assiut University Hospitals, Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed SA, Elhadad AF, Farghaly HS. Evaluation of the effectiveness of valproic acid for treating cyanotic breath holding spells: A Pilot prospective study. Expert Rev Clin Pharmacol. 2020 Nov;13(11):1263-1270. doi: 10.1080/17512433.2020.1828059. Epub 2020 Nov 1. PMID 32969724